CLINICAL TRIAL: NCT02384135
Title: Age-adjusted D-dimer Cutoff Levels to Rule Out Deep Vein Thrombosis: a Prospective Outcome Study
Acronym: ADJUST-DVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: The Ottawa Hospital (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marc Righini, Prof, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-191
Record Dates: First submitted 2015-02-25; First posted 2015-03-10 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Deep Vein Thrombosis; D-dimer
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional (Other): Patients with D-dimer levels between the usual cutoff and the age-adjusted cutoff will be left untreated and followed-up for three months
  Interventions: Other: Three-month thromboembolic risk in patient with D-dimer levels between the usual cut-off and the age-adjusted cut-off

INTERVENTIONS:
Other: Three-month thromboembolic risk in patient with D-dimer levels between the usual cut-off and the age-adjusted cut-off

SUMMARY:
Prospective validation of an age-adjusted D-dimer cut-off to rule out deep vein thrombosis (DVT)

DETAILED DESCRIPTION:
Suspected deep vein thrombosis (DVT) is a frequent clinical problem and remains a diagnostic challenge. The diagnostic approach of DVT relies on sequential diagnostic tests, such as the assessment of clinical probability, plasma D-dimer measurement, and compression ultrasonography (CUS).

Clinical probability has a fair predictive accuracy either evaluated implicitly or by clinical prediction rules and is useful for identifying patients with a low prevalence of DVT who can be usually fully investigated by non invasive tests.

The D-dimer test has been extensively evaluated in the exclusion of DVT, particularly in outpatients. ELISA D-dimer and second-generation latex agglutination (immuno-turbidimetric tests) have a remarkably high sensitivity and have been proved safe first-line tests in association with clinical probability to rule out DVT in outcome studies. The clinical usefulness of D-dimer is defined by the proportion of patients in whom DVT may be ruled out by a normal result and it is determined by the specificity. However, ELISA and second-generation latex agglutination (immuno-turbidimetric tests) tests have a quite limited overall specificity of around 35% to 40%.3 Therefore, many investigators tried to increase the D-dimer thresholds in particular in elderly patients to increase the rate of patients in whom the diagnosis could be excluded by this easy and inexpensive test. Several studies have shown that D-dimer levels increase with age, which turns in a decreased specificity of the D-dimer test at the usual threshold in the elderly, and thus to a less useful test to exclude both DVT and pulmonary embolism (PE) in older patients. For example, ELISA D-dimer is able to rule out PE in 60% of patients aged less than 40 years, but in only 5% of patients above the age of 80. In this study, raising the cutoff value to various points between 600 microg/L and 1000 microg/L increased specificity, but this came at the cost of safety with more false negative test results. In this analysis, however, no stratification was made for clinical probability and the sample was small.

Recently, the investigators retrospectively assessed the value of a progressive cutoff adjusted to age in a wide sample of 1712 patients with suspected PE. This "new" cutoff was defined for D-Dimer test positivity in each patient by multiplying patient's age by 10. All patients with a D-Dimer level below 500 microg/L, and all patients above 50 years whose D-Dimer levels were inferior to their age multiplied by 10 were considered as having a negative D-Dimer test. Using the conventional cutoff, the VIDAS® D-Dimer test was negative (below 500 microg/L) in 512/1712 patients (29.9%) and none had PE during initial workup or the three-month follow-up period.

Using the cutoff adjusted to age (cutoff for D-Dimer test positivity equals age multiplied by ten, in microg/L), the figure was as follows. D-Dimer levels were below the adjusted cutoff in 615/1712 patients (35.9%, number needed to test 2.8). This represented a statistically significant 20.1% increase in the number of patients in whom the D-Dimer test was considered as negative, p=0.0002. Of these 615 patients, 5 had PE during initial workup (0.8%, 95 percent confidence interval 0.4 to 1.9%).

In a recently published a prospective outcome validation study of the age-adjusted cutoff in patients with a clinically suspected PE.13 The study included more than 3300 patients with suspected PE and showed that the three-month thromboembolic risk in patients with an nonhigh (or unlikely) clinical probability and a D-Dimer level between 500 microg/L and the age-adjusted cutoff was of 0.3% (95% CI: 0.1 5 to 1.7%). These results were in line with the one found in patients with a D-dimer level below the usual cutoff of 500 microg/L: 0.1% (95% CI: 0.0% to 0.7%). Moreover, in patients above 75 years the age-adjusted cutoff allowed to increase five-fold the number of patients in whom PE could be excluded without imaging test.

As PE and DVT are often considered as a similar disease, the investigators plan a prospective outcome study in which this progressive or "new" cutoff (age X 10 µg/L) will be used in patients with suspected DVT. In this multicentre study, clinical probability will be assessed by the Wells score (Table 1) and an ELISA D-dimer test (Vidas D-dimer Exclusion® test (Biomérieux, Marcy l'Etoile, Paris, France) or an immuno-turbidimetric test Innovance D-dimer (Siemens, Munich, Germany) will be performed. Patients with a nonhigh or "unlikely" clinical probability with the Wells score and a normal "new" D-dimer cutoff will be considered as not having DVT, and will be followed for three-months to assess possible VTE recurrences. The main outcome will be the rate of thromboembolic events during a formal 3-month follow-up in patients not anticoagulated on the basis of this strategy. Patients with a D-dimer measurement above the age-adjusted cutoff will be investigated with CUS as currently admitted.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients admitted to the emergency ward for suspected DVT will be included in the study, provided they correspond to the following diagnostic and exclusion criteria and they have signed an informed consent form.

Exclusion Criteria:

* DVT suspicion raised more than 48 hours after admission to the hospital
* Pregnancy.
* Patients anticoagulated for a disease other than venous thromboembolism (for instance, atrial fibrillation)
* Concommitant PE suspicion
* Life expectancy less than 3 months
* Absence of informed consent
* Incapacity to deliver informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Three-month thromboembolic risk in patient with D-dimer levels between the usual cut-off and the age-adjusted cut-off | three-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marc Righini, MD, Principal Investigator — University Hospital, Geneva; Grégoire Le Gal, MD, Principal Investigator — Ottawa University Hospital
Locations (15):
- Canada (11):
  - Foothills Medical Centre, Calgary, Calgary/Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - Hôpital Monfort, Monfort, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Providence Health Care, Vancouver, Vancouver/British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa
  - Thunder Bay regional Health Sciences center, Thunder Bay, Ontario
  - University Health network, Toronto, Ontario
- Grégoire LE GAL, Brest, France
- Switzerland (3):
  - Marc Righini, Geneva
  - Geneva University Hospital, Geneva
  - University Hospital of Geneva, Geneva

REFERENCES:
- [Derived] Le Gal G, Robert-Ebadi H, Thiruganasambandamoorthy V, Moustafa F, Penaloza A, Catella J, Grenot MC, Visser S, Mazzolai L, Plumacker A, Barco S, Lang E, Tagalakis V, Deroche C, Garnett M, Hulme J, Roy PM, Ghuysen A, Couturaud F, Engelberger R, El Kouri D, Aujesky D, Righini M; ADJUST-DVT Investigators. Age-Adjusted D-Dimer Cutoff Levels to Rule Out Deep Vein Thrombosis. JAMA. 2026 Jan 5:e2521561. doi: 10.1001/jama.2025.21561. Online ahead of print. PMID 41490105